CLINICAL TRIAL: NCT04487652
Title: Effect of Ubiquinone (Coenzyme Q10) on Early Wound Healing Following Gingival Recession Coverage: a Pilot Study
Brief Title: Ubiquinone (Coenzyme Q10) Application After Gingival Recession Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-01542
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomised placebo-controlled, double blinded, mono-centric trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo spray (Placebo Comparator): Spray consists of matrix out of water, phospholipids and glycerine, plus coloration Colour Sunset Yello E 110 to mimic the test spray
  Interventions: Other: Gingival recession coverage; Drug: with placebo spray application
- CoQ10 spray (Experimental): The CoQ10 spray contains a high quality Kaneka A10 containing CoQ10 trans-isomers which is embedded in a matrix out of water, phospholipids and glycerine. Adana Pharma GmbH is processing the CoQ10 substance into the matrix. One application contains 7 mg CoQ10.
  Interventions: Other: Gingival recession coverage; Drug: with CoQ10 spray application

INTERVENTIONS:
Other: Gingival recession coverage — The Modified Coronally Advanced Tunnel technique in conjunction with a palatal subepithelial connective tissue graft will be performed.
Drug: with CoQ10 spray application — After surgical recession coverage a CoQ10 spray will be applied during the early phase of wound healing.
  Arms: CoQ10 spray
Drug: with placebo spray application — After surgical recession coverage a placebo spray will be applied during the early phase of wound healing.
  Arms: Placebo spray

SUMMARY:
This randomised double blinded clinical trial has the aim to assess the effect of ubiquinone (Coenzyme Q10) on early wound healing following gingival recession coverage. Coenzyme Q10 (CoQ10) is a critical intermediate of the mitochondrial electron transport chain for the synthesis of adenosine triphosphate. The biological importance of CoQ10 is related to antioxidant activity, which can scavenge free radicals as well as restore the antioxidant defence system. Both in vitro and animal studies have suggested that CoQ10 acts as anti-inflammatory agent reducing the inflammatory response by inhibiting the translocation of nuclear factor kappa beta into the nucleus.

Gingival recessions particularly in the esthetic area have become a common indication for treatment. The use of subepithelial palatal connective tissue graft (SCTG) in conjunction with either a coronally advanced flap (CAF) or a coronally advanced tunnel are well established techniques for both the treatment of single and multiple gingival recessions.

Interestingly, despite the fact that CoQ10 is widely investigated, virtually no information exists on its effects upon early wound healing of oral tissues. Therefore, the aim of this study is to investigate the effect of CoQ10 on wound healing after gingival recession surgery.

DETAILED DESCRIPTION:
Gingival recessions constitute a common problem in the adult population worldwide. In the United States the prevalence of ≥1 mm recession in persons >30 years was 58%, representing over 60 million adults while in a French cohort aged 30-65 years old 84.6% had at least one gingival recession. In two other studies it has been reported that over 90% of adults aged 35 to 50 years and above present with single or multiple gingival recessions. The consequences of gingival recessions can be gingivitis due to suboptimal oral hygiene, tooth mobility and in extreme circumstances tooth loss. Tooth sensitivity, root caries, non-carious cervical lesions and esthetic concerns especially with anteriorly located recessions can be also encountered. With the yearly increase in the number of orthodontic patients a potentially additional burden is expected in the population.

The use of subepithelial palatal connective tissue graft (SCTG) in conjunction with either coronally advanced flap (CAF) or coronally advanced tunnel are well established techniques for the treatment of single and multiple gingival recessions. These techniques have been shown to result in predictable root coverage, higher increase in keratinized tissue and stable long-term outcomes thus being considered today state of the art.

Coenzyme Q10 (CoQ10), referred to as 'ubiquinone', is endogenously synthesised by the mevalonate pathway in the human body and is obtained in much of human diet. CoQ10 is a critical intermediate of the mitochondrial electron transport chain for the synthesis of adenosine triphosphate. The biological importance of CoQ10 is related to antioxidant activity, which can scavenge free radicals as well as restore the antioxidant defence system. Furthermore, in vitro and animal studies have suggested that CoQ10 acts as anti-inflammatory agent reducing the inflammatory response by inhibiting the translocation of nuclear factor kappa beta into the nucleus. Owing to its anti-oxidative and anti-inflammatory capacities CoQ10 is of potential therapeutic value in numerous chronic diseases including periodontitis, rheumatoid arthritis or cardiovascular disease. Moreover, it might exert also beneficial effects on wound healing by reducing inflammation and oxidative stress. A recent clinical trial showed that the serum level of TNF-α was significantly reduced in patients with rheumatoid arthritis who received capsules of CoQ10 (100mg/day) for 8 weeks. However, to date, no published study has investigated the anti-oxidative and anti-inflammation effects of coenzyme Q10 spray on oral wound healing. Thus, the purpose of this clinical study is to examine the early wound healing after coenzyme Q10 spray administration (for 3 weeks) in patients undergoing recession coverage surgery.

For this pilot study 30 patients exhibiting single or multiple gingival recessions (Miller class I-III) will randomly be assigned to the control or test group and will be using a placebo or CoQ10 spray for 3 weeks. The primary endpoint is:

• the progress of wound healing assessed by the early wound healing index EHI previously defined by Wachtel et al. 2003.

The secondary endpoints are:

* the improvement of patients' postoperative comfort see patient questionnaire (VAS scale)
* the percentage of root coverage after 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with single and multiple Miller class I, II and III gingival recessions will be included
* Written informed consent

Exclusion Criteria:

* Patients with a history of chronic inflammatory disease
* Patients with severe systemic diseases
* Patients with any sign of clinical infection
* Patients smoking > 5 cigarettes
* Pregnant or lactating women
* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Early wound healing assessed by the early wound healing index by Wachtel | assessed 2 days after surgery
  The early wound healing index by Wachtel describes 5 different stages of wound healing from no fibrin coverage until pus formation.
Early wound healing assessed by the early wound healing index by Wachtel | assessed 7 days after surgery
  The early wound healing index by Wachtel describes 5 different stages of wound healing from no fibrin coverage until pus formation.
Early wound healing assessed by the early wound healing index by Wachtel | assessed 14 days after surgery
  The early wound healing index by Wachtel describes 5 different stages of wound healing from no fibrin coverage until pus formation.
Early wound healing assessed by the early wound healing index by Wachtel | assessed 21 days after surgery
  The early wound healing index by Wachtel describes 5 different stages of wound healing from no fibrin coverage until pus formation.

SECONDARY OUTCOMES:
VAS scale | 2 days until 21 days postoperatively
  The patients'postoperative pain level, 1000 mm scale with 0 representing "no pain" and 1000 mm representing "maximal pain"
Percentage of root coverage | 6 months postoperatively
  How much expressed in percentage of the baseline recession is covered after 6 months
Increase of Keratinized tissue | 6 months postoperatively
  How much keratinized tissue has been gained
Esthetic outcome | 6 months postoperatively
  Esthetic outcomes will be assessed by the root coverage esthetic score, established by Cairo et al. 2009. Parameters like gingival texture, full coverage, marginal tissue contour, scar tissue are evaluated. The maximal score is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Sculean, Prof., Principal Investigator — University of Bern
Locations (1):
- Department of Periodontology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Upon request the individual participant data will be shared

REFERENCES:
- [Background] Lanzrein C, Guldener K, Imber JC, Katsaros C, Stahli A, Sculean A. Treatment of multiple adjacent recessions with the modified coronally advanced tunnel or laterally closed tunnel in conjunction with cross-linked hyaluronic acid and subepithelial connective tissue graft: a report of 15 cases. Quintessence Int. 2020;51(9):710-719. doi: 10.3290/j.qi.a44808. PMID 32577705
- [Background] Guldener K, Lanzrein C, Eliezer M, Katsaros C, Stahli A, Sculean A. Treatment of single mandibular recessions with the modified coronally advanced tunnel or laterally closed tunnel, hyaluronic acid, and subepithelial connective tissue graft: a report of 12 cases. Quintessence Int. 2020;51(6):456-463. doi: 10.3290/j.qi.a44492. PMID 32368762
- [Background] Liu HT, Huang YC, Cheng SB, Huang YT, Lin PT. Effects of coenzyme Q10 supplementation on antioxidant capacity and inflammation in hepatocellular carcinoma patients after surgery: a randomized, placebo-controlled trial. Nutr J. 2016 Oct 6;15(1):85. doi: 10.1186/s12937-016-0205-6. PMID 27716246
- [Background] Sahebkar A, Simental-Mendia LE, Stefanutti C, Pirro M. Supplementation with coenzyme Q10 reduces plasma lipoprotein(a) concentrations but not other lipid indices: A systematic review and meta-analysis. Pharmacol Res. 2016 Mar;105:198-209. doi: 10.1016/j.phrs.2016.01.030. Epub 2016 Feb 2. PMID 26836888
- [Background] Alam MA, Rahman MM. Mitochondrial dysfunction in obesity: potential benefit and mechanism of Co-enzyme Q10 supplementation in metabolic syndrome. J Diabetes Metab Disord. 2014 May 23;13:60. doi: 10.1186/2251-6581-13-60. eCollection 2014. PMID 24932457
- [Result] Stahli A, Imber JC, Raptis E, Salvi GE, Eick S, Sculean A. Effect of enamel matrix derivative on wound healing following gingival recession coverage using the modified coronally advanced tunnel and subepithelial connective tissue graft: a randomised, controlled, clinical study. Clin Oral Investig. 2020 Feb;24(2):1043-1051. doi: 10.1007/s00784-019-03008-6. Epub 2019 Jul 9. PMID 31290017